CLINICAL TRIAL: NCT04245176
Title: Genetic Testing for All Breast Cancer Patients (GET FACTS)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Myriad Genetics, Inc. (Industry)
Responsible Party: Principal Investigator, Tari King, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-509
Record Dates: First submitted 2020-01-17; First posted 2020-01-28 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer; Invasive Breast Cancer; In Situ Breast Cancer; Genetic Testing
Keywords: Breast Cancer; Invasive Breast Cancer; in Situ Breast Cancer; Genetic Testing; Quantitative genetic counseling; Standard genetic counseling
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Quantitative Genetic Counseling (Experimental): The research study procedures include screening for eligibility and study interventions including evaluations and follow up visits - After receiving genetic testing, participants will be placed into one of two counseling methodology groups:
  -- Quantitative genetic counseling: Discussion is guided by tables and graphs.
  Interventions: Behavioral: Quantitative Genetic Counseling
- STANDARD GENETIC COUNSELING (Active Comparator): The research study procedures include screening for eligibility and study interventions including evaluations and follow up visits - After receiving genetic testing, participants will be placed into one of two counseling methodology groups:
  -- Standard genetic counseling: Standard of care discussion
  Interventions: Behavioral: Standard Genetic Counseling

INTERVENTIONS:
Behavioral: Standard Genetic Counseling — Standard genetic counseling: Standard of care discussion
  Arms: STANDARD GENETIC COUNSELING
Behavioral: Quantitative Genetic Counseling — Quantitative genetic counseling: Discussion is guided by tables and graphs.
  Arms: Quantitative Genetic Counseling

SUMMARY:
This study is designed to determine the impact of a novel genetic counseling method on surgical decisions in individuals with newly diagnosed breast cancer

This research study involves an expedited and surgery-specific form of genetic counseling.

The names of the study methods involved in this trial are/is:

* Quantitative genetic counseling (discussion is guided by tables and graphs)
* Standard genetic counseling

DETAILED DESCRIPTION:
* The research study procedures include screening for eligibility and study interventions including evaluations and follow up visits
* After receiving genetic testing, participants will be placed into one of two counseling methodology groups:

  * Standard genetic counseling: Standard of care discussion
  * Quantitative genetic counseling: Discussion is guided by tables and graphs.
* Participants will be on the research study for up to six months, with an optional extension to two years.
* It is expected that about 450 people will participate.
* This research study is a Feasibility Study, which is the first-time investigators are examining this form of genetic counseling.
* This is a randomized study. Randomization means being put into a group by chance. It is like flipping a coin. Neither the participant nor the Investigator will choose the group the participant is assigned to.

ELIGIBILITY:
Inclusion Criteria

* Patients with a new breast cancer diagnosis (invasive or in-situ) considering genetic testing
* Patients with good understanding of written and spoken English
* Patients with apparent cognitive capacity to make surgical decisions for themselves
* Patients who are medically cleared for surgery
* Patients must be at least age 18 but under 79

Exclusion Criteria

* Previous breast cancer diagnosis (invasive or DCIS)
* Metastatic breast cancer
* Patients who have received prior broad-based panel testing (prior BRCA1/2 testing with negative results allowed)
* Bilateral breast cancer
* Known medical or surgical contraindication to contralateral mastectomy
* Hematologic malignancy necessitating skin biopsy/fibroblast culture for germline genetic testing malignancy other than cervical cis or basal or squamous cell skin cancers.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in patient's assessment of their personal contralateral breast cancer risk | 1 month
  A short survey, self-developed in conjunction with the Dana Farber Cancer Institute professional survey core, will be used to compare changes in patients' personal contralateral breast cancer (CBC) risk assessment after quantitative versus standard genetic counseling. The question reads: "By the time you turn 80 years old, what do you believe is the chance you will develop cancer in the other (unaffected) breast?" and answer options are in 10% increments (ie. 0-10%, 11-20%, 21-30%). Their individual assessment of their risk will be collected before and after genetic counseling and will be compared to CBCRisk (for those without gene mutations) or ASK2ME (for those with gene mutations).
Change in patient's propensity to choose bilateral mastectomy as determined by a short self-developed survey question | 1 month
  Patient's will be surveyed about their personal propensity to choose a bilateral mastectomy as the surgical treatment of a unilateral cancer before and after quantitative vs. standard counseling. This survey question was self-developed in conjunction with the Dana Farber Cancer Institute professional survey core. The question reads: "How likely or unlikely are you to choose surgery to remove both breasts (bilateral mastectomy) for your cancer in one breast (unilateral or one-sided breast cancer)?"s answer options include the following: "Very unlikely, Somewhat unlikely, Unsure (neither likely nor unlikely), Somewhat likely, Very likely).

SECONDARY OUTCOMES:
Genetic Testing Satisfaction | 6 Months
  Breast cancer patient satisfaction with genetic counseling practices,comparing the delivery of results by quantitative counseling versus standard counseling, as measured by the Genetic Testing Satisfaction Survey (GTS).
Contralateral Prophylactic Mastectomy (CPM) Rate | 6 Months
  CPM rates will be measured and compared between patients who undergo quantitative versus standard genetic counseling.
Level of anxiety among participants, as measured by the PROMIS anxiety scale | 6 months
  Patients' level of anxiety will be compared between quantitative versus standard genetic counseling to monitor that we are avoiding undue stress on the patients. We will use the Patient-Reported Outcomes Information System (PROMIS) anxiety scale. Scores can range from 8-40, with 40 indicating worse anxiety.
Number of participants with decisional regret (testing and surgery choices) | 6 months
  Decisional regret will be measured and compared between quantitative versus standard genetic counseling, for both the decision to undergo genetic testing and the surgical choice that was made.

CONTACTS AND LOCATIONS:
Overall Officials: Tara King, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Derived] Weiss A, Braun D, Stopfer J, Zhao J, McGrath M, Bradshaw KR, Rosito MS, Davis D, Garber JE, King TA. Genetic Testing for All Breast Cancer Patients: The GET FACTS Randomized Clinical Trial. JAMA Netw Open. 2026 Jan 2;9(1):e2551553. doi: 10.1001/jamanetworkopen.2025.51553. PMID 41525075